CLINICAL TRIAL: NCT01952548
Title: Study Comparing the Pharmacokinetics, Pharmacodynamics, and Safety of K-312 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: K-312-1.01US
Record Dates: First submitted 2013-09-19; First posted 2013-09-30 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Safety and Tolerability

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (14):
- Dose 1 Active (Experimental)
  Interventions: Drug: K-312
- Dose 2 Active (Experimental)
  Interventions: Drug: K-312
- Dose 3 Active (Experimental)
  Interventions: Drug: K-312
- Dose 4 Active (Experimental)
  Interventions: Drug: K-312
- Dose 5 Active (Experimental)
  Interventions: Drug: K-312
- Dose 6 Active (Experimental)
  Interventions: Drug: K-312
- Dose 7 Active (Experimental)
  Interventions: Drug: K-312
- Dose 1 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Dose 2 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Dose 3 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Dose 4 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Dose 5 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Dose 6 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Dose 7 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: K-312
  Arms: Dose 1 Active; Dose 2 Active; Dose 3 Active; Dose 4 Active; Dose 5 Active; Dose 6 Active; Dose 7 Active
Drug: Placebo
  Arms: Dose 1 Placebo; Dose 2 Placebo; Dose 3 Placebo; Dose 4 Placebo; Dose 5 Placebo; Dose 6 Placebo; Dose 7 Placebo

SUMMARY:
This study will test single doses of the study drug in increasing amounts to see if it is safe.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent before any study-specific evaluation is performed.
* Subject is a healthy adult male or a female of non-childbearing potential between the ages of 18 and 45 years, inclusive.
* Subject has a body mass index of 18.5 to 32 kg/m2, inclusive.

Exclusion Criteria:

* Subject is a woman who is of childbearing potential or is breastfeeding.
* Subject has the presence of an active or recurring clinically significant cardiovascular, pulmonary, renal, endocrine, hepatic, neurologic, psychiatric, immunologic, hematologic, gastrointestinal, or metabolic disease requiring medical treatment.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Dates: Start 2013-05; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 10 Days

CONTACTS AND LOCATIONS:
Locations (1):
- Austin, Texas, United States